CLINICAL TRIAL: NCT02717871
Title: Swiss PACK-CXL (Photoactivated Chromophore for Infectious Keratitis Cross-linking) Multicenter Trial for the Treatment of Infectious Keratitis
Brief Title: Swiss PACK-CXL Multicenter Trial for the Treatment of Infectious Keratitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Farhad Hafezi, Professor, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CER 11-198
Record Dates: First submitted 2016-03-09; First posted 2016-03-24 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Keratitis; Infectious Disease (Manifestation)
Keywords: Collagen cross-linking, PACK-CXL, infectious keratitis, CXL.
MeSH Terms: conditions — Keratitis; Communicable Diseases | interventions — Corneal Cross-Linking; Cefazolin; Gentamicins; Pharmaceutical Preparations; Cyclopentolate; Ophthalmic Solutions; Fluoroquinolones; besifloxacin; Ciprofloxacin; Gatifloxacin; Levofloxacin; Moxifloxacin; Ofloxacin; Adrenal Cortex Hormones; prednisolone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (PACK-CXL) (Experimental): Photoactivated chromophore for infectious keratitis-corneal cross-linking (PACK-CXL)
  Interventions: Device: PACK-CXL
- Antimicrobial therapy (Active Comparator): Control arm consists of standard topical antimicrobial therapy recommended for the treatment of microbial keratitis by the American Academy of Ophthalmology.
  Initial empiric topical antibiotic therapy (eye drops or ocular ointment):
  1a. Cefazolin (50mg/ml) in combination with either tobramycin (9-14mg/ml) or gentamicin (9-14mg/ml).
  OR
  1b. a Fluoroquinolones (Besifloxacin 6 mg/ml; ciprofloxacin 3 mg/ml; gatifloxacin 3 mg/ml; levofloxacin 15 mg/ml; moxifloxacin 5 mg/ml; ofloxacin 3 mg/ml)
  2. Cycloplegic agents (cyclopentolate 1% eye drops): to decrease pain and synechia risk is at the physician discretion.
  3. Corticosteroids (prednisolone acetate 0.5% or 1% eye drops): use of corticosteroids for patients included in the study only after complete closure of the epithelium
  Interventions: Drug: Cefazolin in combination with either tobramycin or gentamicin; Drug: Cycloplegic agents (cyclopentolate 1% eye drops); Drug: Fluoroquinolones (Besifloxacin ; ciprofloxacin ; gatifloxacin ; levofloxacin ; moxifloxacin ; ofloxacin ); Drug: Corticosteroids (prednisolone acetate 0.5% or 1% eye drops)

INTERVENTIONS:
Device: PACK-CXL — Local anesthesia
  - Oxybuprocaine or Tetracaine, 1 drop each, applied together, every 3 minutes, total of 3 times
  Abrasio - Abrasio: 1 mm around the borders of the infiltrate/ulcer
  Corneal scrape
  Hypo-osmolaric riboflavin solution
  - Apply one drop every 2 minutes for 20 minutes
  UV-A irradiation
  * 3 mW/cm2 for 30 minutes or 9 mW/cm2 for 10 minutes, 18 mW/cm2 for 5 minutes, 30 mW/cm2 for 3 minutes all allowed (see paper Richoz et al)
  * Treatment diameter: use a irradiation diameter of 6 to 8 mm, keep the infiltrate/ulcus centered.
  Additional postoperative treatment
  * Homatropin or Scopolamin, if anterior chamber reaction
  * Systemic NSAID/NSAR, if substantial pain
  * Do not use: topical or systemic steroids, topical NSAID/NSAR, paracetamol, vitamin A ointment, patching
  Other Names: Corneal cross-linking
  Arms: Treatment (PACK-CXL)
Drug: Cefazolin in combination with either tobramycin or gentamicin — Control arm consists of standard topical antimicrobial therapy recommended for the treatment of microbial keratitis by the American Academy of Ophthalmology.
  Initial empiric topical antibiotic therapy (eye drops or ocular ointment):
  1a. Cefazolin (50mg/ml) in combination with either tobramycin (9-14mg/ml) or gentamicin (9-14mg/ml).
  Other Names: drug
  Arms: Antimicrobial therapy
Drug: Cycloplegic agents (cyclopentolate 1% eye drops) — Cycloplegic agents (cyclopentolate 1% eye drops): to decrease pain and synechia risk is at the physician discretion.
  Arms: Antimicrobial therapy
Drug: Fluoroquinolones (Besifloxacin ; ciprofloxacin ; gatifloxacin ; levofloxacin ; moxifloxacin ; ofloxacin ) — Fluoroquinolones (Besifloxacin 6 mg/ml; ciprofloxacin 3 mg/ml; gatifloxacin 3 mg/ml; levofloxacin 15 mg/ml; moxifloxacin 5 mg/ml; ofloxacin 3 mg/ml)
  Arms: Antimicrobial therapy
Drug: Corticosteroids (prednisolone acetate 0.5% or 1% eye drops) — Corticosteroids (prednisolone acetate 0.5% or 1% eye drops): use of corticosteroids for patients included in the study only after complete closure of the epithelium
  Arms: Antimicrobial therapy

SUMMARY:
To assess the safety and efficacy of PACK-CXL (photoactivated chromophore for infectious keratitis cross-linking) as a firstline treatment for infectious corneal infiltrates and early corneal ulcers, and compare it to the current standard of care, antimicrobial therapy.

DETAILED DESCRIPTION:
Research relevant to this study In 2008, a new concept was taken from transfusion medicine and transferred to ophthalmology: the reduction of pathogen load in platelet concentrates is achieved by treatment of concentrates with riboflavin (Vit B2 as a chromophore and UV-A light). In analogy, a research group in Zurich, Switzerland, showed that this application could be also applied in human corneal infection.

The proof-of-principle study included 5 corneas that were therapy-resistant to any conventional type of treatment. In all five cases, the corneal infection calmed down within days to weeks and all eyes could be saved. In the same year, the effect of riboflavin/UV-A irradiation was shown on several bacteria and fungi in vitro, with a killing rate of almost 98% within 30 minutes for the most common strains responsible for bacterial keratitis like Methicillin resistant Staph aureus and Pseudomonas aeruginosa. A case series and a clinical phase 1 study performed by Makdoumi et al showed the beneficial effect of PACK-CXL (photoactivated chromophore for the treatment of infectious keratitis-corneal collagen crosslinking) in 15 eyes of 15 patients with early onset corneal ulcers. Here, PACK-CXL was even used as the primary therapy, whereas controls received maximal conventional therapy (medication). Again, PACKCXL alone was beneficial in the outcome in all eyes investigated. Between 2010 and 2013, a randomized prospective clinical trial was performed examining the effect of adjuvant PACK-CXL therapy in advanced corneal ulcers with associated melting. Even in these far advanced cases with impending perforation, the additional effect of PACK-CXL was significant, with a drop in the ulcer-related complication rate from 23% (controls) to 0%. A number of smaller reports and case series have shown the effect of PACK-CXL on other bacterial, and also fungal infections.

Study's overall goal The overall goal of this study is to demonstrate that PACK-CXL is not just a valuable adjuvant therapy, but rather a primary treatment modality used in the beginnings of a corneal ulcer, at the stage of an infiltrate or beginning ulcer. Current standard of care would then rather play a secondary, supporting role than a primary one.

Importance of the study on global eye health. The economic and socioeconomic costs related to corneal ulcers and their medical treatment are immense. For example, treatment of a fungal ulcer might cost several thousands of US Dollars. PACK-CXL, in contrast, does not require (expensive) medication, but rather Vitamin B2 solution and a light source. Also, in vitro and in vivo data show that PACK-CXL is highly efficient in antibiotic-resistant infection with MRSA. Furthermore, PACK-CXL is based on CXL, a well-established technique used in other corneal diseases.

Rationale A Riboflavin solution is administered to the cornea in the form of eye drops to the patient. After an administration of 25 minutes (one drop every 2 minutes), the cornea is then irradiated with UV-A light at a wavelength of 365nm and a total energy of 5.4 J/cm2 (use 30 min @ 3 mW/cm2, 10 min @ 9 mw/cm2, or 5 min @ 18mW/cm2). These settings are identical with the standard CXL settings routinely used in clinical practice worldwide. The safety of these settings has been verified in multiple experimental and clinical studies over the past 15 years.

Our hypothesis PACK-CXL might be highly beneficial in the treatment of corneal infection for patients, as an adjuvant therapy in advanced cases, and also a primary mode of treatment in early cases. In this study, the patients are to be examined after treatment with closer control range than is customary at this condition.

The treatment is in clinical use and has a strong theoretical support. Patients will not run an increased risk of injury compared with conventional treatments, as the checks are more frequent than normal and thus, the slightest sign of progress can be detected early. The investigators do not expect any increased suffering from the treatment or inferior healing compared to the usual treatment for patients. The study offers the possibility of a new tool to treat a difficult condition, where the need of culturing decreases and reduces use of antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Patient exhibit clinical signs of corneal infiltrate or beginning corneal ulcer on at least one eye, of suspected bacterial, fungal or mixed (bacterial and fungal) origin.
* Infiltrates and early ulcers up to a maximum 2mm in diameter; may lie close to the corneal limbus, but at a minimal distance of 2mm from central cornea.
* Infiltrates and early ulcer depth of a maximum of 300 μm, assessed by either OCT or Scheimpflug imaging
* All lesions must show an open epithelium with fluorescein positive staining
* No previous antibiotic/antifungal treatment OR at least no antibiotic/antifungal treatment for a minimum of 48 hours from last treatment
* Provide signed and dated patient consent form
* Patient willing to comply with all study procedures and be available for the duration of the study
* Male or female, >18 years of age. No children or adolescents of 18 years and less of age will be included in this study.

Exclusion Criteria:

* Lesion/infiltrate involving the central 2mm diameter of the cornea
* Suspicion of non-infectious keratitis, viral or acanthamoeba keratitis or sterile infiltrate.
* Closed epithelium over the lesion
* Pachymetry of less than 400 microns at the thinnest point.
* Patients who cannot participate in the treatment or be monitored with frequent clinician controls as required in the study protocol.
* Corneal perforation
* Descemetocele
* Pregnancy or breastfeeding
* Active corneal herpetic disease
* Systemic treatment involving steroids
* Immunosuppressed/immune-compromised patients
* Patients with diagnosed eczema (or atopic dermatitis)
* Previous keratoplasty
* Patients with monocular vision

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-03; Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Time to re-epithelialization of the corneal surface | 28 days

SECONDARY OUTCOMES:
Time from treatment to discharge of the patient | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Hafezi, MD, PhD, Principal Investigator — fhafezi@elza-institute.com
Locations (1):
- University of Geneva, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goldstein MH, Kowalski RP, Gordon YJ. Emerging fluoroquinolone resistance in bacterial keratitis: a 5-year review. Ophthalmology. 1999 Jul;106(7):1313-8. PMID 10406613
- [Background] Whitcher JP, Srinivasan M, Upadhyay MP. Corneal blindness: a global perspective. Bull World Health Organ. 2001;79(3):214-21. Epub 2003 Jul 7. PMID 11285665
- [Background] Goodrich RP. The use of riboflavin for the inactivation of pathogens in blood products. Vox Sang. 2000;78 Suppl 2:211-5. PMID 10938955
- [Background] Iseli HP, Thiel MA, Hafezi F, Kampmeier J, Seiler T. Ultraviolet A/riboflavin corneal cross-linking for infectious keratitis associated with corneal melts. Cornea. 2008 Jun;27(5):590-4. doi: 10.1097/ICO.0b013e318169d698. PMID 18520510
- [Background] Martins SA, Combs JC, Noguera G, Camacho W, Wittmann P, Walther R, Cano M, Dick J, Behrens A. Antimicrobial efficacy of riboflavin/UVA combination (365 nm) in vitro for bacterial and fungal isolates: a potential new treatment for infectious keratitis. Invest Ophthalmol Vis Sci. 2008 Aug;49(8):3402-8. doi: 10.1167/iovs.07-1592. Epub 2008 Apr 11. PMID 18408193
- [Background] Schrier A, Greebel G, Attia H, Trokel S, Smith EF. In vitro antimicrobial efficacy of riboflavin and ultraviolet light on Staphylococcus aureus, methicillin-resistant Staphylococcus aureus, and Pseudomonas aeruginosa. J Refract Surg. 2009 Sep;25(9):S799-802. doi: 10.3928/1081597X-20090813-07. Epub 2009 Sep 11. PMID 19772254
- [Background] Makdoumi K, Mortensen J, Crafoord S. Infectious keratitis treated with corneal crosslinking. Cornea. 2010 Dec;29(12):1353-8. doi: 10.1097/ICO.0b013e3181d2de91. PMID 21102196
- [Background] Makdoumi K, Mortensen J, Sorkhabi O, Malmvall BE, Crafoord S. UVA-riboflavin photochemical therapy of bacterial keratitis: a pilot study. Graefes Arch Clin Exp Ophthalmol. 2012 Jan;250(1):95-102. doi: 10.1007/s00417-011-1754-1. Epub 2011 Aug 27. PMID 21874347
- [Background] Moren H, Malmsjo M, Mortensen J, Ohrstrom A. Riboflavin and ultraviolet a collagen crosslinking of the cornea for the treatment of keratitis. Cornea. 2010 Jan;29(1):102-4. doi: 10.1097/ICO.0b013e31819c4e43. PMID 19730094
- [Background] Pot SA, Gallhofer NS, Matheis FL, Voelter-Ratson K, Hafezi F, Spiess BM. Corneal collagen cross-linking as treatment for infectious and noninfectious corneal melting in cats and dogs: results of a prospective, nonrandomized, controlled trial. Vet Ophthalmol. 2014 Jul;17(4):250-60. doi: 10.1111/vop.12090. Epub 2013 Aug 14. PMID 23941330
- [Derived] Hafezi F, Hosny M, Shetty R, Knyazer B, Chen S, Wang Q, Hashemi H, Torres-Netto EA; PACK-CXL Working Group. PACK-CXL vs. antimicrobial therapy for bacterial, fungal, and mixed infectious keratitis: a prospective randomized phase 3 trial. Eye Vis (Lond). 2022 Jan 7;9(1):2. doi: 10.1186/s40662-021-00272-0. PMID 34996516
- [Derived] Davis SA, Bovelle R, Han G, Kwagyan J. Corneal collagen cross-linking for bacterial infectious keratitis. Cochrane Database Syst Rev. 2020 Jun 17;6(6):CD013001. doi: 10.1002/14651858.CD013001.pub2. PMID 32557558